CLINICAL TRIAL: NCT05244941
Title: Remote By Default 2: The New Normal
Brief Title: Remote By Default 2: Optimising the Remote-by-default Model in the United Kingdom (UK) General Practice
Acronym: RBD2
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Oxford (Other)
Collaborators: University of Plymouth (Other); Nuffield Trust (Unknown)
Responsible Party: Sponsor
Other Study IDs: 300719
Record Dates: First submitted 2021-10-27; First posted 2022-02-17 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cross site-case study: Qualitative methods: semi-structured interviews for patients, front line clinical practitioners, and health system stakeholders, case study building across sites

SUMMARY:
Aim; To inform high-quality, safe and equitable care in the United Kingdom (UK) general practice (GP) in the context of policies which require phone, video or e-consultation by default.

BACKGROUND When COVID struck, general practice shifted to predominantly phone, video or e-consultations instead of face-to-face. Remote had benefits (e.g. reducing spread of COVID), but also downsides (technical glitches; inequalities of access; missed diagnoses; reduced continuity of care; and patients simply not seeking care at all). Despite this, the Secretary of State for Health of the UK, Matt Hancock declared on 30th July 2020 that remote-by-default is here to stay.

RESEARCH QUESTION To what extent is remote-by-default, introduced for infection control during the pandemic, fit for purpose for the long term - and how can we make remote care better and safer?

DESIGN AND METHODS Mixed-method case study with co-design workshops and cross-sector stakeholder events.

OBJECTIVES AND METHODS

1. GP PRACTICES The investigators will support 10 GP practices to develop effective remote services and alternatives where needed. The investigators will help them collect data and use their findings to inform improvement efforts.
2. PATIENTS The investigators will interview 40 patients selected for diversity (age, ethnicity, locality, socio-economic status, condition[s], digital literacy), and hold two workshops (one remotely and one in person, Covid allowing) where patients help co-design ways to combine remote and face-to-face models.
3. WIDER SYSTEM The investigators will engage stakeholders - including policymakers, professional bodies, industry, civil society and patient groups - in ongoing dialogue about how to deliver and support a more equitable, less risky remote-by-default service. The investigators will interview patients and hold cross-sector stakeholder events (big Zoom meetings), working both before and after the events to build relationships and action ideas.

DETAILED DESCRIPTION:
AIM: To inform a more fit-for-purpose remote-by-default model in UK general practice which takes account of a) quality and safety of care, b) equity and inclusivity, c) staff wellbeing and training, and d) the wider technical and regulatory infrastructure.

STRATEGIC OBJECTIVES

1. PRACTICE LEVEL: Follow a sample of 10 GP practices for two years as they seek to introduce, improve and sustain remote-by-default consultations, supporting practices in developing effective remote services and equitable alternatives to remote where needed.
2. PATIENT LEVEL: Capture the patient experience of remote-by-default consultations and ensure that this perspective is incorporated in practice- and system-level efforts to improve and augment remote-by-default services.
3. SYSTEM LEVEL: Engage a wide range of stakeholders - including policymakers, the UKs National Health Service (NHS), professional bodies, industry, civil society and patient groups - in an ongoing dialogue about how to deliver and support a more equitable, less risky remote-by-default service.

OPERATIONAL OBJECTIVES

1. PRACTICE LEVEL:

   1. Using an embedded researcher-in-residence model, build relationships with 10 GP practices selected for maximum variety in digital maturity, geographic location (e.g. urban/rural/remote) and population demographics. Support patient and public involvement (PPI) reps in those practices.
   2. Undertake interviews (up to 10 per practice) and collect documentary data (e.g. protocols, patient leaflets, workload data) from each practice to build a case study.
   3. Follow practice case studies longitudinally over time, supporting them to a) optimise quality and safety of care; b) ensure digital inclusion and provide equitable alternatives for the digitally excluded; c) maintain wellbeing and train and support their staff; d) overcome infrastructural hurdles (both technical and regulatory).
   4. Run two online co-design workshops for up to 40 people each (with hands-on activities in small groups), incorporating insights from patient/carer workshops (see below).
2. PATIENT LEVEL:

   1. Recruit a diverse sample of 40 service users (patients and carers), most of whom will be registered with participating GP practices, with some identified through patient groups or snowballing, ensuring that the investigators include a range of people at risk of digital exclusion.
   2. Through narrative interviews (by phone, video or face to face as preferred), capture the patient/carer experience of remote-by-default consultations across four key quality and safety areas (long term condition monitoring, getting an appointment with own clinician, symptoms that could indicate early cancer, and complex multi-morbidity).
   3. Hold two co-design workshops (one remote and one face to face), each with up to 20 patients and carers, to generate insights about how digital inclusion impacts on access and quality and safety of care, and generate a range of 'digital inclusion personas'.
3. SYSTEM LEVEL:

   1. Build relationships with key stakeholders (listed under strategic objective 3) through up to 30 elite interviews and extending our ongoing stakeholder map.
   2. Hold four large, cross-sector stakeholder events, including preparatory and follow-up activities, focused respectively on quality and safety of care; digital inclusion (informed by digital inclusion personas); staff wellbeing, training and supervision; and technical and regulatory infrastructure.

METHODS Mixed-method, multi-site case study with co-design workshops and cross-sector stakeholder events. 'Mixed methods', is defined as, "research in which … researchers combine elements of qualitative and quantitative approaches … for the broad purposes of breadth and depth of understanding and corroboration".

DELIVERABLES Range of patient/carer experience of remote, 4 digital inclusion workshops, support for change in 10 GP practices, cross-case learning, 4 cross-sector stakeholder events with follow-on support for policy action, academic papers and policy briefings, lay summaries and resources.

ELIGIBILITY:
Inclusion Criteria:

* over 18
* willing and able to provide informed consent
* diagnosed with any relevant condition, receiving care from participating services

Exclusion Criteria:

* inability to read or speak English unless a relevant translator is available
* co-morbidity preventing participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General population
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Qualitative experience of remote by default care access in the primary care setting in the UK | through study completion, an average of 2 years
  Iteratively develop support for change in 10 GP practices to inform a more fit for purpose model of remote by default care access in the primary care setting in the UK
Support for cross stakeholder policy action on informing a fit for purpose remote by default care access in the primary care setting in the UK | through study completion, an average of 2 years
  Support for cross stakeholder policy action, through creation of policy briefs, academic papers and resources

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oxford, Oxford, United Kingdom